CLINICAL TRIAL: NCT03571490
Title: Improving Postoperative Pain Management With the Ultrasound-guided Transmuscular Quadratus Lumborum Block for Elective Laparoscopic Hand-assisted Nephrectomy and Robot-assisted Partiel Nephrectomy: A Double Blind, Randomized, Placebo Controlled Trial
Brief Title: Ultrasound-guided Transmuscular Quadratus Lumborum Block for Elective Laparoscopic Hand-assisted Nephrectomy and Robot Assisted Partiel Nephrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: V2.02.05.2017; 2017-002130-23 (EudraCT Number)
Record Dates: First submitted 2017-10-27; First posted 2018-06-27 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Pain; Ultrasound Guided Transmuscular Quadratus Lumborum Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TQL Ropivacaine(active) (Active Comparator): Bilateral Single shot of ropivacaine 0.325% 30 mL. In total 60 mL of 0.325% ropivacaine
  Interventions: Drug: Ropivacaine
- TQL saline (placebo) (Placebo Comparator): Bilateral single shot of saline 0.9% 30 mL. in Total 60 mL of saline 0.9%
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — Single shot of ropivacaine 0.325%
  Arms: TQL Ropivacaine(active)
Drug: Saline — Single shot of saline 0.9%
  Arms: TQL saline (placebo)

SUMMARY:
Patients with kidney cancer often undergo hand-assisted laparoscopic nephrectomy or Robot assisted partiel nephrectomy. The investigators performed a one-year retrospective study. the sudy revealed that 67% of the patients needed substantial amounts of opioids for postoperative pain management (PPM) in recovery despite a multimodal analgesic regime. In a prospective pilot study including ten laparoscopic hand-assisted nephrectomy, with severe postoperative pain the investigators found that bilateral Ultrasound-guided (USG) transmuscular quadratus lumborum (TQL) block substantially reduced pain and opioid consumption. This study aims to evaluate the effect on PPM of a bilateral USG TQL block compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* Kidney cancer
* Have received thorough information, orally and in written
* Signed the "Informed Consent" form on participation in the trial

Exclusion Criteria:

* Inability to cooperate
* Inability to speak and understand Danish both orally and written
* Allergy to local anaesthetics or opioids
* Daily intake of opioids
* Local infection at the site of injection or systemic infection
* Difficulty visualisation of muscular and fascial structures in ultrasound visualisation necessary to the block administration
* Known abuse of alcohol or medicine
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 12 hours postoperatively
  Opioid consumption postoperatively: data from Patient Controlled Analgesia(PCA) pump and patient medical record).

SECONDARY OUTCOMES:
opioid consumption | 6 hours postoperatively
  Opioid consumption postoperatively (data from PCA pump and patient medical record).
opioid consumption | 18 hours postoperatively
  Opioid consumption postoperatively (data from PCA pump and patient medical record).
opioid consumption | 24 hours postoperatively
  Opioid consumption postoperatively (data from PCA pump and patient medical record).
NRS score | 12 hours postoperatively
  Numeric Rating Scale(NRS). Scores range from 0-10, 0=no pain-10=worst pain postoperatively at rest and activity
NRS score at rest and activity | 6 hours postoperatively
  Numeric Rating Scale(NRS). Scores range from 0-10, 0=no pain-10=worst pain
NRS score at rest and activity | 18 hours postoperatively
  Numeric Rating Scale(NRS). Scores range from 0-10, 0=no pain-10=worst pain
NRS score at rest and activity | 24 hours postoperatively
  Numeric Rating Scale(NRS). Scores range from 0-10, 0=no pain-10=worst pain
Opioid-related side effects | 6 hours postoperatively
  The degree of morphine-related side effects (PONV, itching, fatigue, etc.)
Opioid-related side effects | 12 hours postoperatively
  The degree of morphine-related side effects (PONV, itching, fatigue, etc.)
Opioid-related side effects | 18 hours postoperatively
  The degree of morphine-related side effects (PONV, itching, fatigue, etc.)
Opioid-related side effects | 24 hours postoperatively
  The degree of morphine-related side effects (PONV, itching, fatigue, etc.)
Patient satisfaction with application of the block. NRS | Immediately after application of the block
  Numeric Rating Scale(NRS). Scores range from 0-10, 0=no pain-10=worst pain
Ambulation | within 24 hours postoperatively
  Time from operation to ambulation

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand university Hospital, Anaesthesiology, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dam M, Hansen C, Poulsen TD, Azawi NH, Laier GH, Wolmarans M, Chan V, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block reduces opioid consumption and prolongs time to first opioid demand after laparoscopic nephrectomy. Reg Anesth Pain Med. 2021 Jan;46(1):18-24. doi: 10.1136/rapm-2020-101745. Epub 2020 Oct 26. PMID 33106280